CLINICAL TRIAL: NCT02932696
Title: Post Infarction Exercise Training Effects on Systolic and Diastolic Myocardial Function Assessed by 2D Strain Ultrasound
Brief Title: Post Infarction Exercise Effects on Myocardial Function Assessed by 2D Strain Ultrasound
Acronym: TrainStrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIMAO/2016-06/AD-01
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): Patients in this arm were encouraged to participate in an exercise training program, and they accepted to do so.
  Intervention: Cardiac training program
  Interventions: Other: Cardiac training program
- No exercise training (No Intervention): Patients in this arm were encouraged to participate in an exercise training program, and they refused to do so.

INTERVENTIONS:
Other: Cardiac training program — This program takes place at the Cardiovascular Rehabilitation Department at the Nîmes University Hospital and includes a combination of various physical activities: treadmill, exercise bike, rower, aerobics, gymnastics, serious games, swimming. The program begins approximately within 3 months after myocardial infarction and consists of 20 consecutive days of training. The main physical activity is aerobic interval training (AIT).
  30-minute AIT sessions will occur 5x per week for 4 weeks.
  1 AIT session includes a warm up for 8 minutes to reach a heart rate during exercise corresponding to 20 to 30% of maximum aerobic power determined during the initial effort test. Then interval training occurs with 4x2 min of high intensity effort (heart rate during exercise corresponding to 80% of maximum aerobic power) alternating with 2 min of active recovery at 20-30% of maximum aerobic power. Then recovery for 8 minutes.
  Arms: Exercise training

SUMMARY:
The main goal of our project is to study and describe the effect of exercise training on systolic and diastolic myocardial function assessed by 2D ultrasound strain after myocardial infarction.

Our working hypothesis is that the intrinsic myocardial contractility and relaxation assessed by global longitudinal strain in phase II (or 2D strain) during post-infarction exercise training will be improved compared to baseline values as well as compared to values in a no-training group. Should this hypothesis prove true, it would help explain the improvements in functional capacity observed during the post-infarction period and after exercise training.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 4 months of follow-up
* The patient had a first myocardial infarction episode (within the past 3 months) requiring medical treatment or revascularisation (e.g. balloon angioplasty) or aortocoronary bypass

Exclusion Criteria:

* The patient is simultaneously participating in (or has participated in the past 3 months) another interventional study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection or under guardianship
* It is impossible to correctly inform the patient or the patient refuses to sign the consent
* The patient is pregnant, parturient, or breastfeeding
* Contra indication for exercise training
* Valve prosthesis
* Severe valvular disease
* Pacemaker
* Heart transplant
* Non sinus rhythm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
The % global longitudinal strain of the left ventricle | within 3 months post infarction = T0 (baseline)
The % global longitudinal strain of the left ventricle | 5 weeks
The % global longitudinal strain of the left ventricle | 3 months

SECONDARY OUTCOMES:
maximal oxygen consumption (VO2max; mL/min/kg) | within 3 months post infarction = T0 (baseline)
maximal oxygen consumption (VO2max; mL/min/kg) | T0 + 5 weeks
maximal oxygen consumption (VO2max; mL/min/kg) | T0 + 3 months
maximum aerobic power (watts) | within 3 months post infarction = T0 (baseline)
maximum aerobic power (watts) | T0 + 5 weeks
maximum aerobic power (watts) | T0 + 3 months
First ventilatory threshold (mL/min/kg) | within 3 months post infarction = T0 (baseline)
First ventilatory threshold (mL/min/kg) | T0 + 5 weeks
First ventilatory threshold (mL/min/kg) | T0 + 3 months
left ventricle longitudinal systolic strain rate | within 3 months post infarction = T0 (baseline)
left ventricle longitudinal systolic strain rate | T0 + 5 weeks
left ventricle longitudinal systolic strain rate | T0 + 3 months
left ventricle longitudinal diastolic strain rate | within 3 months post infarction = T0 (baseline)
left ventricle longitudinal diastolic strain rate | T0 + 5 weeks
left ventricle longitudinal diastolic strain rate | T0 + 3 months
% radial systolic strain | within 3 months post infarction = T0 (baseline)
% radial systolic strain | T0 + 5 weeks
% radial systolic strain | T0 + 3 months
% radial diastolic strain | within 3 months post infarction = T0 (baseline)
% radial diastolic strain | T0 + 5 weeks
% radial diastolic strain | T0 + 3 months
% circumferential systolic strain | within 3 months post infarction = T0 (baseline)
% circumferential systolic strain | T0 + 5 weeks
% circumferential systolic strain | T0 + 3 months
% circumferential diastolic strain | within 3 months post infarction = T0 (baseline)
% circumferential diastolic strain | T0 + 5 weeks
% circumferential diastolic strain | T0 + 3 months
Radial systolic strain rate | within 3 months post infarction = T0 (baseline)
Radial systolic strain rate | T0 + 5 weeks
Radial systolic strain rate | T0 + 3 months
Radial diastolic strain rate | within 3 months post infarction = T0 (baseline)
Radial diastolic strain rate | T0 + 5 weeks
Radial diastolic strain rate | T0 + 3 months
Circumferential systolic strain rate | within 3 months post infarction = T0 (baseline)
Circumferential systolic strain rate | T0 + 5 weeks
Circumferential systolic strain rate | T0 + 3 months
Circumferential diastolic strain rate | within 3 months post infarction = T0 (baseline)
Circumferential diastolic strain rate | T0 + 5 weeks
Circumferential diastolic strain rate | T0 + 3 months
Telediastolic volume (mL) | within 3 months post infarction = T0 (baseline)
Telesystolic volume (mL) | T0 + 5 weeks
Telesystolic volume (mL) | T0 + 3 months
Telediastolic volume (mL) | T0 + 5 weeks
Telediastolic volume (mL) | T0 + 3 months
Left ventricle mass (g/m^2) | within 3 months post infarction = T0 (baseline)
Left ventricle mass (g/m^2) | T0 + 5 weeks
Left ventricle mass (g/m^2) | T0 + 3 months
Ejection fraction of the left ventricle | within 3 months post infarction = T0 (baseline)
Ejection fraction of the left ventricle | T0 + 5 weeks
Ejection fraction of the left ventricle | T0 + 3 months
S' wave velocity (cm/s) | within 3 months post infarction = T0 (baseline)
S' wave velocity (cm/s) | T0 + 5 weeks
S' wave velocity (cm/s) | T0 + 3 months
E' wave velocity (cm/s) | within 3 months post infarction = T0 (baseline)
E' wave velocity (cm/s) | T0 + 5 weeks
E' wave velocity (cm/s) | T0 + 3 months
A' wave velocity (cm/s) | within 3 months post infarction = T0 (baseline)
A' wave velocity (cm/s) | T0 + 5 weeks
A' wave velocity (cm/s) | T0 + 3 months
The E/A ratio | within 3 months post infarction = T0 (baseline)
The E/A ratio | T0 + 5 weeks
The E/A ratio | T0 + 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France